CLINICAL TRIAL: NCT03149939
Title: Use of Febuxostat in Hyperuricemia Among Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Collaborators: New Jeddah Clinic Hospital (Industry)
Responsible Party: Principal Investigator, Mahmoud Hamada imam, MD. - Lecturer at Internal Medicine Department- Faculty of Medicine, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN-0316
Record Dates: First submitted 2017-05-10; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Hyperuricemia; Hemodialysis Complication
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Febuxostat 40 milligramsTablet — Febuxostat 40 milligramsTablet every other day for 3 months

SUMMARY:
Hyperuricemia is not infrequently encountered among hemodialysis patients. However, there is no clear data about use of febuxostat among hemodialysis patients, apart from very small case series. The aim of this study is to investigate the efficacy of using febuxostat for the treatment of Hyperuricemia among hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Hemodialysis patient
* Hyperuricemia (Uric acid level above 6.0 mg/dL in females and 7.0 mg/dL in males)

Exclusion Criteria:

* Patient currently and/or recently received drugs for hyperuricemia within the last three months
* Patient had recent (within 3 months) change of erythropoiesis stimulating drugs or other drug known to increase uric acid e.g furosemide

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Change in serum uric acid | at three months of Febuxostat 40 milligrams Tablet therapy
  Change in serum uric acid after 3 months of Febuxostat 40 milligrams Tablet therapy

IPD SHARING:
Plan to Share IPD: No